CLINICAL TRIAL: NCT03412097
Title: Assessing New or Worsening Symptoms (Aka Adverse Events for This Study) After Chiropractic Care at a Chiropractic Teaching Clinic: An Active Surveillance Pilot Study
Brief Title: (MIST1)-Part 1: Assessment & Feasibility of Post-Symptoms Evaluation
Acronym: MIST1
Status: Completed | Type: Observational
Sponsor: Parker University (Other)
Collaborators: University of Texas at Tyler (Other); University of Alberta (Other); Canadian Memorial Chiropractic College (Other)
Responsible Party: Sponsor
Other Study IDs: Parker16_001
Record Dates: First submitted 2018-01-17; First posted 2018-01-26 (Actual); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Patient Safety; Manipulation, Spinal
Keywords: chiropractic; SMT; active surveillance reporting system
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: active surveillance — Provides a structure to systematically gather adverse event information from healthcare providers and sometimes directly from patients.

SUMMARY:
To increase patient safety culture in spinal manipulation therapy (SMT) this study will assess the ability to implement an active surveillance reporting system for a chiropractic teaching clinic and determining preliminary incidence of adverse events (AE) following SMT performed by the chiropractic interns. Adverse events defined for the primary outcome of this study is any new or worsening symptom following a chiropractic encounter.

DETAILED DESCRIPTION:
Healthcare systems acknowledge the importance of patient safety including the reduction of preventable adverse events (AE). For healthcare providers who perform spinal manipulation therapy (SMT), the investigation of AEs remains in its infancy for several reasons including finding a reporting system that accurately collects AEs information, varied descriptions of AE's severity and occurrence frequency and the variable natural history of musculoskeletal conditions treated by SMT. Together, these factors act together to conspire against the implementation of systematic changes in SMT application that would result in improved patient care and safety.

In addition, it is vital that patient safety training initiates at the start of a healthcare worker's career. This pilot active surveillance study was designed to assess the feasibility of collecting data on patients' self-report of symptom changes as well as interns' report at a chiropractic teaching clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the Parker University Wellness Clinic
* Agreed to participate

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive Patients
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Pohlman, DC, MS, PhD, Principal Investigator — Parker University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who agreed to participate in the study completed a pretreatment form. After treatment, patients were asked to complete a post-treatment form. Complete information was received on 89 patients (pretreatment and post-treatment forms).
Groups:
- Consecutive Patients: Data from consecutive patients who sought care at Parker University's teaching clinic.
Period: Overall Study
Arm/Group | Consecutive Patients
Started | 89
Completed | 89
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients who agreed to participate in the study (364 encounters) completed a pretreatment form. After treatment, patients were asked to complete a post-treatment form. Complete information was received on 89 unique patients (pretreatment and post-treatment forms) totaling 119 patient encounters.
Groups:
- Consecutive Patients: Patients who agreed to participate in the study (364 encounters) completed a pretreatment form. After treatment, patients were asked to complete a post-treatment form. Complete information was received on 89 unique patients (pretreatment and post-treatment forms) totaling 119 patient encounters.
Arm/Group | Consecutive Patients
Number analyzed (Participants) | 89
Age, Continuous [Mean (Full Range); unit: years] | 39.5 [1 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Patient Encounters That Report a New or Worsening Symptom
Description: An adverse advent is any unfavorable sign, symptom or disease temporarily associated with the treatment, whether or not caused by the treatment, specifically any worsened or new symptom reported by the patient up to one week after care.
Time Frame: Up to 7 days post treatment - Day 0-7
Population: 89 patients completed both the pre and post-treatment forms received. These were considered complete and thus used for study analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Consecutive Patients
Number analyzed (Participants) | 89
Participants | 8

ADVERSE EVENTS:
Time Frame: 0-7 days
Description: 1. All-Cause Mortality
  2. Serious Adverse Events
  3. Other (Not Including Serious) Adverse Events - This study's primary outcome definition for an adverse event is any unfavorable sign, symptom or disease temporarily associated with the treatment, whether or not caused by the treatment, specifically any worsened or new symptom reported by the patient up to one week after care.
Groups:
- All Consecutive Patients: Patients who agreed to participate in the study (consecutive) completed a pretreatment form. After treatment, patients were asked to complete a post-treatment form. Complete information was received on 89 patients (pretreatment and post-treatment forms).
Arm/Group | All Consecutive Patients
All-Cause Mortality (participants affected / at risk) | 0/89
Serious Adverse Events (participants affected / at risk) | 0/89
Other Adverse Events (participants affected / at risk) | 8/89
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Consecutive Patients (N=89)
Worsening or new symptom (Musculoskeletal and connective tissue disorders) | 8 — Worsened and new symptoms were considered AEs (adverse events).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No